CLINICAL TRIAL: NCT06010810
Title: The Effectiveness of 3% Topical Tranexamic Acid Compared to 4% Topical Hydroquinone as Therapy of Melasma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nevi Yasnova, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23040463
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 % Topical Tranexamic Acid (Experimental): Patients will receive 3% Topical Tranexamic Acid, on half of the face, twice a day for a total duration of 2 months
  Interventions: Drug: 3 % Topical Tranexamic Acid
- 4 % Topical Hydroquinone (Experimental): Patients will receive 4% Topical Hydroquinone, on half of the face, twice a day for a total duration of 2 months.
  Interventions: Drug: 4% Topical Hidroquinone

INTERVENTIONS:
Drug: 3 % Topical Tranexamic Acid — Patient will be given 3% Topical Tranexamic Acid, on half of the face, twice a day for 2 months
  Arms: 3 % Topical Tranexamic Acid
Drug: 4% Topical Hidroquinone — Patient will be given 4% Topical Hidroquinone, on half of the face, twice a day for 2 months
  Arms: 4 % Topical Hydroquinone

SUMMARY:
The goal of this clinical trial is to compare 3% Topical Tranexamic Acid with 4% Topical Hydroquinone as Therapy of Melasma in Patients with Skin Type III-V. The main question[s] it aims to answer are:

1. Is there a greater decrease in mMASI score after application of 3% topical tranexamic acid compared to 4% hydroquinone in melasma patients with skin type III - V?
2. Is there a greater decrease in mexameter score after application of 3% topical tranexamic acid compared to 4% hydroquinone in melasma patients with skin type III - V?
3. Are there any side effects of topical therapy of 3% tranexamic acid cream on melasma patients with skin types III - V? Participants with melasma diagnostic will apply the tranexamic acid cream and hydroquinone cream on both sides of the face differently. Researchers will compare by measuring the mexameter score and mMasi score to see if there any decrease in both sides of the face.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with melasma.
* 18-60 years old.
* Fitzpatrick skin type III to V.
* Willing to be a research subject (SP) and sign a consent sheet. research (informed consent).

Exclusion Criteria:

* Are pregnant and/or breastfeeding
* History of taking hormonal contraceptives in the last 6 months
* History of topical melasma therapy: corticosteroids, tretinoin, hydroquinone, and Another therapy that lightens the skin in the last 2 weeks.
* Use oral systemic therapy or injection in melasma, such as oral acid tranexamic, oral antioxidant, vitamin C injection, and glutathione injection in 4 last week.
* History of superficial peeling therapy in the last 4 weeks.
* History of deep peeling, laser or mechanical abrasion therapy in the last 6 months.
* Use drugs that are photosensitizers such as phenytoin, tetracycline, spironolactone, and carbamazepine.
* History of bleeding disorders or being on blood-thinning therapy
* Allergy to tranexamic acid
* Difficulty in complying with treatment.
* Are experiencing symptoms of COVID-19, such as fever, cough, sore throat, loss of sense of taste or smell, red eyes, diarrhea, rash on the skin

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified Melasma Area and Severity Index | 2 months
  Decrease of Modified Melasma Area and Severity Index
Mexameter score | 2 months
  Decrease of melanin index and erythema index

CONTACTS AND LOCATIONS:
Overall Officials: Nevi Yasnova, MD, Principal Investigator — Faculty of medicine, University of Indonesia
Locations (1):
- Cipto Mangungkusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El-Husseiny R, Rakha N, Sallam M. Efficacy and safety of tranexamic acid 5% cream vs hydroquinone 4% cream in treating melasma: A split-face comparative clinical, histopathological, and antera 3D camera study. Dermatol Ther. 2020 Nov;33(6):e14240. doi: 10.1111/dth.14240. Epub 2020 Sep 14. PMID 32856757
- [Result] Atefi N, Dalvand B, Ghassemi M, Mehran G, Heydarian A. Therapeutic Effects of Topical Tranexamic Acid in Comparison with Hydroquinone in Treatment of Women with Melasma. Dermatol Ther (Heidelb). 2017 Sep;7(3):417-424. doi: 10.1007/s13555-017-0195-0. Epub 2017 Jul 26. PMID 28748406